CLINICAL TRIAL: NCT06723782
Title: Surgical Release of Hand Tendons with Wrapping of the Released Tendon Using an Amniotic Membrane
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMTRIX-Tenolyse-TBF; 2023-A01189-36 (Other: IDRCB)
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Tendon Adhesion; Tenolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AMTRIX-D (Experimental): Surgical release of the tendon and wrapping of the released tendon with desiccated amniotic membrane (AMTRIX-D)
  Interventions: Biological: AMTRIX-D

INTERVENTIONS:
Biological: AMTRIX-D — Use of a decellularized, viro-inactivated, desiccated, and sterile allogeneic amniotic membrane graft to wrap a tendon after release of its adhesions.

SUMMARY:
The goal of this clinical trial is to evaluate whether an amniotic membrane can function as an effective anti-adhesive barrier following surgical release of tendon adhesions. The main question the clinical trial aims to answer is:

- Can wrapping an amniotic membrane around a surgically released tendon help reduce recurrence of adhesions and promote recovery of hand functionality?

Participants will:

* Undergo surgical treatment (surgical release of the tendon adhesions and wrapping of the amniotic membrane around the release tendon) on Day 0.
* Visit the center for a series of tests 15 days, 6 weeks, 3 months, 6 months after the surgical intervention.

DETAILED DESCRIPTION:
Tendon adhesions are a common problem in hand injuries and can have multiple causes. They can occur as a result of tendon damage itself or in the absence of such damage, following a fracture, crush injury, or infection. During healing, tendons become surrounded by an inflammatory exudate rich in fibrin, which can later turn into scar tissue. This scar tissue forms a strong bond between the tendon and the surrounding tissue, leading to significant functional impairment.

In their epidemiological study of 5,229 flexor tendon repairs, Dy et al. determined that 6% of patients who had undergone primary repair required a second intervention, with surgical release of adhesions around the tendons in 58% of cases. In flexor tendon repairs, adhesions are particularly promoted by damage to the tendon sheath, poor junction of the two severed ends of a lacerated tendon, or ischemia of the tendon and immobilization. Regardless of the etiology, adhesions prevent the efficient gliding of the tendon within its sheath, resulting in a discrepancy between near-normal passive range of motion and limited active range of motion.

When the range of motion deficit persists despite 6 months of high-quality rehabilitation, surgical treatment is considered. Tenolysis and early mobilization are the standard treatments for symptomatic tendon adhesions in the hand. Tenolysis involves surgically releasing the adhesions formed around the tendons. Follow-up rehabilitation after tendon surgical release can help reduce adhesion formation, though it does not completely prevent their formation or recurrence after tenolysis.

In recent years, many strategies have been proposed to limit adhesion formation after tendon repair surgery in the hand, or recurrence after tenolysis. Tested physical barriers include, among others, the interposition of an amniotic membrane or a composite of hyaluronic acid and methylcellulose, local application of sodium hyaluronate or various gels derived from proteoglycans or hyaluronan, or the use of non-steroidal anti-inflammatory drugs.

However, no definitive solution has yet been found, and to date, the use of anti-adhesion barriers remains limited in routine practice.

The product developed by TBF is set in this context with the goal of offering a safe biological solution that would minimize adhesion recurrence after tenolysis and promote the recovery of hand functionality.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 to 65 years old
* Adhesion of a flexor and/or extensor tendon of the hand.
* Adhesion localized to a single finger.
* Adhesion that has been present for at least 3 months following primary repair, despite high-quality rehabilitation. Primary repair is defined as the repair of a tendon injury, fracture, crush injury of the finger, infection, etc., leading to the adhesion of the tendon to surrounding tissue.
* Patient with a total passive range of motion of the proximal and distal interphalangeal joints of at least 150°.
* Informed and consenting patient.
* Patient enrolled in a social security plan or a beneficiary of such a plan.

Exclusion Criteria:

* Pregnant or breastfeeding woman, or without an effective method of contraception.
* Patient requiring tenolysis after tendon grafting for the reconstruction of a deep common flexor or after reimplantation.
* Patient with amputated hand(s).
* Patient with an untreated fracture or non-union in the affected hand.
* Patient requiring multiple surgical interventions that may be potential confounding factors, particularly those involving additional incisions.
* Patient unable to understand rehabilitation or follow the study protocol.
* Patient with a contraindication to anesthesia.
* Person deprived of liberty by judicial or administrative decision.
* Adult subject to legal protection measures or incapable of expressing consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in the finger total active range of motion | 6 months
  Total active range of motion of the finger evaluated according to Strickland's classification: (TAM/175) × 100, where TAM = flexion of the proximal interphalangeal joint + flexion of the distal interphalangeal joint - extension deficit. Total active range of motion scores are expressed as percentages and classified into four categories: poor if < 25%, moderate from 25% to 49%, good from 50% to 74%, and excellent if > 75%. The primary objective of the study will be achieved if the total active range of motion is good or excellent (>50%) at 6 months.

SECONDARY OUTCOMES:
Change in the daily functionality of the finger | 15 days, 6 weeks, 3 months, 6 months
  Daily functionality of the finger evaluated using Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire (0 = no disability, 100 = most severe disability).
Change in finger pain | 15 days, 6 weeks, 3 months, 6 months
  Pain evaluated from 0 (no pain) to 10 (worst imaginable pain) on a visual analog scale (VAS).
Change in hand grip strength | 6 weeks, 3 months, 6 months
  Grip strength measured in kg by grip strength test using a hand dynamometer.
Frequency of occurrence of post-surgical complications | 15 days, 6 weeks, 3 months, 6 months
  Evaluation of the frequency of occurrence of post-surgical complications and in particular rupture of the deep common flexor tendon, phlegmon, wound dehiscence.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Chirurgical de la Main et du Membre Supérieur, Lyon, France

IPD SHARING:
Plan to Share IPD: No